CLINICAL TRIAL: NCT00850772
Title: Early Post-Operative Enteral Feeding in Patients With Advanced Epithelial Ovarian Cancer
Acronym: OPEN
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Queensland Centre for Gynaecological Cancer (Other Government)
Collaborators: Cancer Australia Priority-driven Collaborative Cancer Research Scheme (Unknown); The University of Queensland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: OPEN
Record Dates: First submitted 2009-02-23; First posted 2009-02-25 (Estimated); Last update posted 2014-06-12 (Estimated); Status verified 2014-06

CONDITIONS: Epithelial Ovarian Cancer; Peritoneal Cancer; Fallopian Tube Cancer
Keywords: Enteral nutrition; Ovarian cancer; Peritoneal cancer; Fallopian tube cancer; Malnutrition; Surgery; Gynecological Cancer; Suspected advanced epithelial ovarian cancer
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial; Fallopian Tube Neoplasms; Ovarian Neoplasms; Malnutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Early post-operative enteral feeding (Experimental): Standard post-operative care and diet together with early post-operative enteral feeding
  Interventions: Dietary Supplement: Early post-operative enteral feeding
- Standard post-operative care and diet (No Intervention): Standard post-operative care and diet only

INTERVENTIONS:
Dietary Supplement: Early post-operative enteral feeding — During primary surgical treatment an enteral feeding tube will be inserted through the patient's nose into their small bowel. Enteral feeding will commence 4 hours following return to ward from surgery. Feeding will start at a rate of 40 ml/hr for the first 24 hours, and then increased to goal weight. Goal will be calculated by 125 kiloJoules/kilogram adjusted body weight.
  Arms: Early post-operative enteral feeding

SUMMARY:
Ovarian cancer patients are often at risk of malnutrition because of weight loss, lack of appetite and reduced food intake. Being malnourished can contribute to the incidence and severity of cancer treatment side effects and increase the risk of infection. Currently patients with advanced ovarian cancer do not receive early nutrition using a feeding tube.

The purpose of this study is to compare enteral nutrition along with standard post-surgery care against current standard post-operative care alone. This study will see if early nutrition using a feeding tube has an impact on length of hospital admission, recovery from surgery, complications from surgery, nutritional status and ultimately a reduction in treatment costs in people with Advanced Epithelial Ovarian Cancer (EOC). Primary Peritoneal Cancer (PPC) or Fallopian Tube Cancer. Nutritional support has been shown to ;

* Prevent and treat under-nutrition,
* Enhance anti-tumour treatment effects,
* Reduce adverse effects of anti-tumour therapies,
* Improve quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Patients requiring planned primary surgery for suspected or histologically proven advanced ovarian, primary peritoneal cancer or fallopian tube cancer.
* Signs of moderate or severe malnutrition - Patient Generated Subjective Global Assessment (PG-SGA) Category B or C and/or a total numerical score of 4 or more in the PG-SGA
* Medically fit for primary surgery
* Signed written informed consent
* Females aged 18 years or older

Exclusion Criteria:

* Other histological type than ovarian cancer, peritoneal cancer or fallopian tube cancer
* Recurrent ovarian cancer, peritoneal or fallopian tube cancer
* Pre-existing contraindications to enteral nutrition such as ileus, gastrointestinal ischemia, bilious or persistent vomiting, or mechanical obstruction
* Positive urine pregnancy test
* Unfit for surgery; serious concomitant systemic disorders incompatible with the study (at the discretion of the investigator)
* Participation in other clinical trials that may have an impact on the outcomes of this trial.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2009-01; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Cost outcomes as represented by length of stay and cost effectiveness of enteral feeding / Quality of life | End of study
  Compare treatment costs and cost effectiveness between early enteral feeding with standard post-operative care versus current standard ost-operative care for advanced epithelial ovarian cancer.
  Compare quality of life after surgery between women who receive early enteral feeding along with standard post-operative care versus those who receive current standard post-operative care for advanced epithelial ovarian cancer

SECONDARY OUTCOMES:
length of stay | Until discharge from hospital
  Length of stay in an intensive care unit or high dependency unit and overall length of hospital stay.
Need for inotropic medications and intravenous treatment requirements | Until discharge from hospital
Nutritional status 6 weeks after surgery | 6 weeks after surgery
Treatment related adverse events | End of study
Delay and dose reductions of chemotherapy / quality of life during chemotherapy | End of study

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Obermair, MD FRANZCOG CGO, Study Chair — Queensland Centre for Gynaecological Cancer
Locations (6):
- Australia (6):
  - The Wesley Hospital, Auchenflower, Queensland
  - Brisbane Private Hospital, Brisbane, Queensland
  - Greenslopes Private Hospital, Greenslopes, Queensland
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - Mater Health Services, South Brisbane, Queensland
  - Gold Coast Hospital, Southport, Queensland

REFERENCES:
- [Derived] Baker J, Janda M, Graves N, Bauer J, Banks M, Garrett A, Chetty N, Crandon AJ, Land R, Nascimento M, Nicklin JL, Perrin LC, Obermair A. Quality of life after early enteral feeding versus standard care for proven or suspected advanced epithelial ovarian cancer: Results from a randomised trial. Gynecol Oncol. 2015 Jun;137(3):516-22. doi: 10.1016/j.ygyno.2015.03.048. Epub 2015 Mar 28. PMID 25827292